CLINICAL TRIAL: NCT03928236
Title: Benzodiazepine-free Cardiac Anesthesia for Reduction of Postoperative Delirium
Acronym: B-Free
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B-Free.2019
Record Dates: First submitted 2019-04-18; First posted 2019-04-26 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Delirium; Post-cardiac Surgery
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: Multicenter, cluster-randomized, crossover trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Limited Benzodiazepine Policy (Experimental): Policy of no routine use of any intraoperative benzodiazepines.
  Interventions: Other: Limited Intraoperative Benzodiazepine
- Liberal Benzodiazepine Policy (Active Comparator): Policy for the administration of benzodiazepine as per clinical guidelines but no lower than 0.03 mg/kg (ideal body weight midazolam equivalent) to all patients undergoing cardiac surgery. Any benzodiazepine may be used.
  Interventions: Other: Liberal Intraoperative Benzodiazepine

INTERVENTIONS:
Other: Limited Intraoperative Benzodiazepine — policy for limited use of intraoperative benzodiazepine
  Arms: Limited Benzodiazepine Policy
Other: Liberal Intraoperative Benzodiazepine — policy for liberal use of intraoperative benzodiazepine
  Arms: Liberal Benzodiazepine Policy

SUMMARY:
B-FREE is a pragmatic, multicentre, cluster crossover trial evaluating whether a policy limiting the use of intra-operative benzodiazepine reduces post-operative delirium when compared with a policy of 'ad libitum' administration. The knowledge generated by this study will provide the basis for cardiac anesthesia practice guidelines.

DETAILED DESCRIPTION:
Delirium, an acute state of confusion, occurs in approximately 1 in 5 adults after open heart surgery. Even though it is a temporary state, patients who experience delirium are at increased risk of serious problems that last after the delirium has resolved. These problems include decreases in thinking, mobility, self-care, and the ability to live independently in a community setting. Patients who experience delirium have longer stays in hospital, are more likely to be discharged to a nursing home, and are more likely to die. Benzodiazepines are a sedative and amnestic medication that may be associated with delirium. As such, benzodiazepines are rarely used for sedation in the intensive care unit after cardiac surgery. However, benzodiazepines continue to be used frequently in the operating room by anesthesiologists during open heart surgery because of their amnestic effects and limited impact on blood pressure. Nevertheless, practice is divided among cardiac anesthesiologists, with some never using benzodiazepines and others using them for nearly all patients.

Because the best approach (routine benzodiazepines or restricted benzodiazepines) remains uncertain, we will compare the effect of a hospital policy of intraoperative medication use that includes benzodiazepines to a policy that uses alternative medications and no benzodiazepines on the incidence of delirium after open heart surgery. The findings of the study have the potential to improve the outcomes of tens of thousands of patients around the world and will provide the basis for cardiac anesthesiology practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Hospital is a major surgical center with a minimum of 250 cases of cardiac surgery per year.
* Equipoise by the hospital physicians regarding the use of benzodiazepines during surgery (≥ 95% of hospital cardiac anesthesia group agrees to manage adult patients (age >18 years) as per the benzodiazepine policy in place during a given crossover period).
* Hospital routinely assesses patients (age >18 years) for postoperative delirium at least once every 12 hours during the initial 72 hours after cardiac surgery as a part of routine clinical care using either the Confusion Assessment Method-ICU (CAM-ICU) or the Intensive Care Delirium Screening Checklist (ICDSC).

Exclusion Criteria:

- Hospital does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15886 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Delirium | up to 72 hours post cardiac surgery
  Delirium assessed up to 72 hours after surgery using standardized and validated delirium scales

SECONDARY OUTCOMES:
Number of Days in ICU after Cardiac Surgery | through study completion, approximately 37 months
  Length of Stay (LOS) in Intensive Care Unit after Cardiac Surgery
Number of Days in Hospital after Cardiac Surgery | through study completion, approximately 37 months
  Length of Stay (LOS) in Hospital after Cardiac Surgery
Incidence of In-hospital Mortality | through study completion, approximately 37 months
  Death from any cause after index cardiac surgery and during the index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Spence, MD FRCPC, Principal Investigator — Population Health Research Institute; Eric Jacobsohn, MBChB MPHE, Principal Investigator — University of Manitoba; Stuart Connolly, MD FRCPC, Study Chair — Population Health Research Institute
Locations (20):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Cornell Medicine, New York, New York
- Canada (18):
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hôpital Laval, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Regina General Hospital, Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spence J, Devereaux PJ, Lee SF, D'Aragon F, Avidan MS, Whitlock RP, Mazer CD, Rousseau-Saine N, Rajamohan RR, Pryor KO, Klein R, Tan E, Cameron MJ, Di Sante E, DeBorba E, Mustard ME, Couture EJ, Zamper RPC, Law MWY, Djaiani G, Saha T, Choi S, Hedlin P, Pikaluk DR, Lam W, Deschamps A, Ramasundarahettige CF, Vincent J, McIntyre WF, Oczkowski SJW, Dulong BJ, Beaver C, Kloppenburg SA, Lamy A, Jacobsohn E, Belley-Cote EP; B-Free Investigators and the Canadian Perioperative Anesthesia Clinical Trials Group. Benzodiazepine-Free Cardiac Anesthesia for Reduction of Postoperative Delirium: A Cluster Randomized Crossover Trial. JAMA Surg. 2025 Mar 1;160(3):286-294. doi: 10.1001/jamasurg.2024.6602. PMID 39878960
- [Derived] Spence J, Belley-Cote E, Jacobsohn E, Lee SF, D'Aragon F, Avidan M, Mazer CD, Rousseau-Saine N, Rajamohan R, Pryor K, Klein R, Tan EC, Cameron M, Di Sante E, DeBorba E, Mustard M, Couture E, Zamper R, Law M, Djaiani G, Saha T, Choi S, Hedlin P, Pikaluk R, Lam WY, Deschamps A, Whitlock R, Dulong B, Devereaux PJ, Beaver C, Kloppenburg S, Oczkowski S, McIntyre WF, McFarling M, Lamy A, Vincent J, Connolly S; B-Free Investigators. Benzodiazepine-Free Cardiac Anesthesia for Reduction of Postoperative Delirium (B-Free): A Protocol for a Multi-centre Randomized Cluster Crossover Trial. CJC Open. 2023 Jun 8;5(9):691-699. doi: 10.1016/j.cjco.2023.06.001. eCollection 2023 Sep. PMID 37744662
- [Derived] Wang ML, Min J, Sands LP, Leung JM; the Perioperative Medicine Research Group. Midazolam Premedication Immediately Before Surgery Is Not Associated With Early Postoperative Delirium. Anesth Analg. 2021 Sep 1;133(3):765-771. doi: 10.1213/ANE.0000000000005482. PMID 33721875